CLINICAL TRIAL: NCT01393860
Title: Aliskiren Use in Diabetic Patients: Who's Using it, Why, and How is it Working ?
Brief Title: Real-world Aliskiren Use in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Clinical Disclosure Office, Novartis Pharmaceuticals
Other Study IDs: HEORUS0081
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes; Hypertension
Keywords: Diabetes; aliskiren; hypertension; renal impairment
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Aliskiren: Diabetic nephropathy

SUMMARY:
The purpose of this study is to evaluate real-world patterns of aliskiren use with a focus of change in renal function following aliskiren initiation as well as to identify "triggering events" that lead to aliskiren initiation.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Patients ages 18 yeras and older
* Hypertension Diagnosis
* Currently on at least 1 hypertensive medication
* At least 2 lab measure before and after aliskiren initiation

Exclusion Criteria:

* Inadequate chart records where microalbuminuria, serum creatinine and blood pressure data are not within 3-12 months prior to initiation of Aliskiren
* Pregnancy
* Development of secondary renal disease unrelated to diabetes (such as nephritis)
* Terminal illness
* AIDS/HIV Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with hypertension who were initiated on aliskiren
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Measure: Change in blood pressure | baseline and 1 year

SECONDARY OUTCOMES:
Measure: Change in urine microalbumin | baseline and 1 year
Measure: Change in creatinine | baseline and 1 year
Measure: Change in potassium levels | baseline and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Phamaceuticals
Locations (1):
- MODEL Clinical Research, Research Division of Bay Endocrinology Associates GBMC Physicians pavilion North, Baltimore, Maryland, United States